CLINICAL TRIAL: NCT01658163
Title: Use of 2 Octyl-cyanoacrylate Together With a Self-adhering Mesh for Skin Closure Following Abdominoplasty: An Open, Prospective, Controlled, Randomized Clinical Study
Brief Title: Use of 2-octyl-cyanoacrylate Together With a Self-adhering Mesh
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Prineo
Record Dates: First submitted 2012-05-09; First posted 2012-08-06 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Surgical Wound Dehiscence; Cutis Laxa; Wound of Skin
Keywords: abdominoplasty,; skin closure, dressings
MeSH Terms: conditions — Surgical Wound Dehiscence; Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators prospectively studied the results of wound closure after abdominoplasty with randomized use of PrineoTM and conventional suturing to assess the possible difference in outcome between these two methods.Follow-up visits to the outpatient clinic were scheduled at 2 weeks, 6 months and 12 months after surgery. A panel consisting of three plastic surgeons and three plastic surgery residents assessed the wound and scar appearance during the three follow-up visits.

DETAILED DESCRIPTION:
Abdominoplasty is one of the most commonly performed procedures in plastic surgery. The appearance of the scar is a major factor contributing to the aesthetic outcome of the procedure and depends largely on the technique of wound closure. The new PrineoTM wound closure system was introduced to combine the effectiveness of 2-octyl-cyanoacrylate (Dermabond TM) together with a self-adhering mesh.Fifty-two women and 8 men aged between 21 and 65 years scheduled for abdominoplasty were included in the study. Total operating time after abdominoplasty between the traditional wound closure technique and the PrineoTM-type wound closure technique was compared. Two weeks postoperatively, the wounds were examined and graded according to the Hollander Cosmesis Scale. At 6- and 12-month follow-up, the aesthetic outcome of the abdominal scar was evaluated with the Vancouver Scar Scale. Twelve months postoperatively, the patients were further asked to score their part of the Patient Scar Assessment Scale.There was a statistically significant shorter mean of total operating time for the new skin closure system compared with intradermal sutures. The Hollander Cosmesis Scale indicated a significantly more favourable overall result with PrineoTM at 2 weeks after surgery. The Vancouver Scar Scale demonstrated a better cosmetic outcome in favour of PrineoTM 6 and 12 months after surgery The Patient Scar Assessment Scale scores 12 months after surgery indicated that the patients noted significantly less pain, thickness and irregularity with PrineoTM.Based on our results, we conclude that PrineoTM is a safe and effective substitute for superficial skin closure, with good cosmetic results and no increase in wound complications. The use of PrineoTM decreases operative times and costs and enhances patients' postoperative comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an abdominoplasty without exclusion criteria

Exclusion Criteria:

* current intake of systemic steroids
* known HIV-positive or other immunocompromised status
* known or suspected allergy or sensitivity to cyanoacrylate, formaldehyde, tapes or adhesives
* personal or family history of keloid or hypertrophic scar formation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-06; Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryousch Parvizi, MD, Principal Investigator — Medical University of Graz